CLINICAL TRIAL: NCT06227923
Title: Development and Validation of a Protected Discharge Model Using Technology in Multimorbidity and Poly-treated Older Subjects. The PRO-HOME Study
Brief Title: A Protected Discharge Model Using Technology in Multimorbid and Poly-treated Older Subjects
Acronym: PRO-HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alberto Pilotto (Other)
Responsible Party: Sponsor-Investigator, Alberto Pilotto, Director of Department of Geriatric Care, Orthogeriatrics and Rehabilitation, Ente Ospedaliero Ospedali Galliera
Organization: Ente Ospedaliero Ospedali Galliera (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NET-2016-02361805-1
Record Dates: First submitted 2023-12-22; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Multimorbid and Poly-treated Older People

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants are transferred from the hospital ward to a small apartment with a technological assessment and monitoring established inside the hospital setting.
  Interventions: Device: PRO-HOME intervention
- Control group (No Intervention): Participants remain in the hospital ward and receive normal clinical practice.

INTERVENTIONS:
Device: PRO-HOME intervention — Patients are transferred to the apartment inside the hospital setting and are evaluated and assessed also using technological devices
  Arms: Intervention group

SUMMARY:
The main goal of thi clinical trial is to evaluate if a protected discharge model can reduce the length of hospital stay in older participants aged over 65 years old who have been admitted to the hospital for an acute event and have been considered stable and dischargeable. Participants of the intervention group will be asked to transfer to a small apartment, inside the hospital setting, equipped by technological devices and to be involved in cognitive and physical activities during the stay. Researchers will compare this intervention group with a control group who receive normal clinical practice where older people remain in the hospital ward.

DETAILED DESCRIPTION:
Participants who fit the inclusion criteria are randomized in two arms (intervention or control groups). All of them are evaluated with a comprehensive geriatric assessment (Multidimensional Prognostic Index), a depression scale (Geriatric Depression Scale), quality of Life scale (Short-Form 12 items), and physical parameters (Hand Grip, Short Physical Performance Battery, gait speed). In the intervention group the following clinical parameters will be collected through technological devices: spontaneous physical performance, sleep monitoring, gait speed, quality of movements, heart rate, SpO2, and other vital parameters.

ELIGIBILITY:
Inclusion Criteria:

1. participants aged 65 years or older;
2. admitted to the acute geriatric units for an acute event;
3. deemed stable and dischargeable from the hospital;
4. good personal autonomy in the Activities of Daily Living (ADL) (according to the Katz ADL scoring≥ 3/6);
5. normal cognition or mild cognitive impairment (Short Portable Mental Status Questionnaire (SPMSQ) ≤ 5/10);
6. signed informed consent

Exclusion Criteria:

1. participants aged less than 65 years old
2. not considerable stable and dischargeable
3. ADL <3/6
4. SPMSQ > 5/10
5. not signed informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | At 1 month after the baseline
  Evaluate the efficacy of a protected discharge model in terms of length of hospital stay in multimorbid and poly-treated older subjects

SECONDARY OUTCOMES:
Negative clinical outcome: re-hospitalization | 1, 3 , 6 months after the baseline
  Evaluate negative clinical outcome about re-hospitalization recording the number of re-hospitalization (number of access in the hospital's wards and related reason) related to each patient after the intervention if relevant
Negative clinical outcome: institutionalization | 1, 3 , 6 months after the baseline
  Evaluate negative clinical outcome about institutionalization recording the access in institution related to each patient after the intervention, if relevant
Negative clinical outcome: mortality | 1, 3 , 6 months after the baseline
  Evaluate negative clinical outcome about mortality collecting the data about mortality (date and reason of death) if relevant
Step mean through smartwatch | At baseline
  Units of measure: number of steps
Heart rate through smartwatch | At baseline
  Units of measure: bpm
Daily inactivity time through smartwatch | At baseline
  Units of measure: percentage of time spent inactive
Distance covered through smartwatch | At Baseline
  Units of measure: cm
Gait speed through kinect Azure | At baseline
  Units of measure:meters/second
Trunk/head oscillation (body sway /lean in) through kinect Azure | At baseline
  Units of measure: degrees

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Pilotto, Principal Investigator — EO Galliera
Locations (1):
- EO Ospedali Galliera, Genova, Italy

IPD SHARING:
Plan to Share IPD: No
Results will be published in one or more different papers with only statistically significant data with the description of statistical methods of the analyses.

REFERENCES:
- [Background] Pilotto A, Volta E, Barbagelata M, Argusti A, Camurri A, Casiddu N, Berutti-Bergotto C, Custodero C, Cella A. The PRO-HOME Project. A multicomponent intervention for the protected discharge from the hospital of multimorbid and polytreated older individuals by using innovative technologies: A pilot study. Health Expect. 2024 Feb;27(1):e13872. doi: 10.1111/hex.13872. Epub 2023 Oct 27. PMID 37890856
- [Background] Pilotto A, Barbagelata M, Morganti W, Seminerio E, Iaccarino G, Genazzani A, Trompetto C, Arabia G, Illario M, Volta E, Custodero C, Cella A; MULTIPLAT_AGE Investigators. Development and implementation of multicomponent homecare interventions for multimorbid and frail older people based on Information and Communication Technologies: The MULTIPLAT_AGE project. Arch Gerontol Geriatr. 2024 Feb;117:105252. doi: 10.1016/j.archger.2023.105252. Epub 2023 Nov 3. PMID 37972433
- [Derived] Pilotto A, Morganti W, Barbagelata M, Seminerio E, Morelli S, Custureri R, Dini S, Senesi B, Prete C, Puleo G, Berutti Bergotto C, Vallone F, Custodero C, Camurri A; PRO-HOME Project Investigators Group. A transitional care program in a technologically monitored in-hospital facility reduces the length of hospital stay and improves multidimensional frailty in older patients: a Randomized Clinical Trial. Aging Clin Exp Res. 2024 Aug 6;36(1):160. doi: 10.1007/s40520-024-02821-8. PMID 39105934